CLINICAL TRIAL: NCT02957305
Title: Comparison Between 400 µg or 200 µg of Misoprostol for Cervical Dilatation in 1st Trimester Miscarriage - A Clinical Trial
Brief Title: Misoprostol 400 µg Versus 200 µg for Cervical Ripening in 1st Trimester Miscarriage
Acronym: MISO200
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Ricardo Francalacci Savaris, Head of the Gynecologic Emergency Unit, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160309
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Miscarriage in First Trimester
Keywords: misoprostol; miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, operators and statistical analysis were performed blindly.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol 400 µg (Active Comparator): Participants received misoprostol 400 µg: 2 tablets of misoprostol (200µg each) introduced into the vagina, at least 6 hours before the Manual Vacuum Aspiration (MVA) procedure.
  Interventions: Drug: Misoprostol 400mcg Tab
- Misoprostol 200 µg (Experimental): Participants received misoprostol 200 µg: 1 tablet of misoprostol introduced into the vagina, at least 6 hours before the Manual Vacuum Aspiration procedure.
  Interventions: Drug: Misoprostol 200mcg Tab

INTERVENTIONS:
Drug: Misoprostol 400mcg Tab — 400µg of misoprostol (2 tablets)
  Other Names: Misoprostol control
  Arms: Misoprostol 400 µg
Drug: Misoprostol 200mcg Tab — 200µg of misoprostol (1 tablet)
  Other Names: Misoprostol comparator
  Arms: Misoprostol 200 µg

SUMMARY:
Local current protocol for cervical ripening in 1st trimester miscarriage recommends 400 µg of misoprostol intravaginally 3 hours before uterine evacuation. This regime has been recommended by some international guidelines . So far, there are no recent studies comparing cervical dilatation between 400 µg of misoprostol and a reduced dose (e.g., 200 µg) for 6 hours. If cervical ripening is similar between these two regimens(i.e., 200µg regimen is not inferior to 400µg regimen), costs reductions and lower side effects may be issued without losing quality of cervix dilatation.

DETAILED DESCRIPTION:
Miscarriage is defined by the World Health Organization as the interruption of the pregnancy up to 20-23 weeks, or the products of pregnancy weighing less than 500 grams (1). Nearly 15% of known pregnancies end in miscarriage, especially in the first 12 weeks. Estimates indicate that 68000 women die worldwide each year, as a result of unsafe abortions. Abortions are the major cause of maternal death, particularly in Latin America and the Caribbean. In cases of retained and incomplete abortions, uterine emptying is recommended. In the first trimester of pregnancy, either pharmacological or surgical procedure is accepted according to international guidelines.

Pharmacological treatment for uterine evacuation includes the administration of mifepristone and misoprostol or misoprostol alone. Nevertheless, surgical methods have been shown a greater acceptability and patient satisfaction due to a reduced incidence of adverse effects. Currently, Manual Vacuum Aspiration (MVA) is the technique recommended by the Brazilian Ministry of Health and the Brazilian Federation of Gynecology and Obstetrics.

MVA should be performed after cervical ripening. This pre-surgical procedure makes the procedure safer and more effective. In Brazil, misoprostol is the most suitable drug to be used in these cases because of its efficacy, ease of use, low cost, stability at room temperature, and availability. Misoprostol is a synthetic prostaglandin E1 analog and can be administered by oral, sublingual, buccal, rectal, and vaginal routes.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted at the Gynecological emergency Unit at Hospital de Clínicas de Porto Alegre scheduled for uterine evacuation with <12 weeks of gestation.

Exclusion Criteria:

* patients who do not wish to participate in the project;
* patients with ectopic pregnancy;
* patients with comorbidities (heart failure congestive, chronic obstructive pulmonary disease);
* patients with hypovolemic shock;
* patients with cervical incompetence;
* patients with infected miscarriage/abortion (presence of fever, pus from the cervix, leukocytosis [> 14000]);
* patients with twin pregnancy;
* patients with Marfan syndrome;
* patients allergic to misoprostol;
* patients with coagulopathy;
* patients with opening of cervical internal os (4 mm of dilatation at the time of consultation);
* patients with previous surgery of the cervix (conization);
* patients with concomitant use of IUDs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Ricardo, MD, PhD, Principal Investigator — HCPA
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We intend to share raw data with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: unlimited
Access Criteria: free to read
URL: https://docs.google.com/spreadsheets/d/1WmVYj6LDAHrOqiCaAlq4TmHg8lhFxoucxqewNfOVVkE/edit?usp=sharing

REFERENCES:
- [Background] Kapp N, Lohr PA, Ngo TD, Hayes JL. Cervical preparation for first trimester surgical abortion. Cochrane Database Syst Rev. 2010 Feb 17;2010(2):CD007207. doi: 10.1002/14651858.CD007207.pub2. PMID 20166091
- [Background] Blanchard K, Clark S, Winikoff B, Gaines G, Kabani G, Shannon C. Misoprostol for women's health: a review. Obstet Gynecol. 2002 Feb;99(2):316-32. doi: 10.1016/s0029-7844(01)01701-x. PMID 11814515
- [Background] Marret H, Simon E, Beucher G, Dreyfus M, Gaudineau A, Vayssiere C, Lesavre M, Pluchon M, Winer N, Fernandez H, Aubert J, Bejan-Angoulvant T, Jonville-Bera AP, Clouqueur E, Houfflin-Debarge V, Garrigue A, Pierre F; College national des gynecologues obstetriciens francais. Overview and expert assessment of off-label use of misoprostol in obstetrics and gynaecology: review and report by the College national des gynecologues obstetriciens francais. Eur J Obstet Gynecol Reprod Biol. 2015 Apr;187:80-4. doi: 10.1016/j.ejogrb.2015.01.018. Epub 2015 Jan 31. PMID 25701235
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Ectopic Pregnancy and Miscarriage: Diagnosis and Initial Management in Early Pregnancy of Ectopic Pregnancy and Miscarriage. London: RCOG Press; 2012 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK132775/ PMID 23638497
- [Background] ACOG Committee Opinion. American College of Obstetrician and Gynecologist. ACOG Committee Opinion. Number 283, May 2003. New U.S. Food and Drug Administration labeling on Cytotec (misoprostol) use and pregnancy. Obstet Gynecol. 2003 May;101(5 Pt 1):1049-50. doi: 10.1016/s0029-7844(03)00396-x. PMID 12738178
- [Background] Tang J, Kapp N, Dragoman M, de Souza JP. WHO recommendations for misoprostol use for obstetric and gynecologic indications. Int J Gynaecol Obstet. 2013 May;121(2):186-9. doi: 10.1016/j.ijgo.2012.12.009. Epub 2013 Feb 19. PMID 23433680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diagnosis of miscarriage and scheduled for Manual Vacuum Aspiration at the Gynecologic Emergency Unit of Hospital de Clínicas de Porto Alegre, a tertiary teaching hospital, were recruited. The first participant was enrolled on December 21, 2016.
Pre-assignment Details: A total of 269 were screened. From these, 211 were enrolled and randomized to treatment. After randomization, 2 cases, one case of infected abortion and one case with previous cervical conization were identified and they were treated as for intention to treat.
Groups:
- Misoprostol 400µg: Participants received misoprostol 400 µg: 2 tablets of misoprostol (200µg each) were introduced into the vagina, at least 6 hours before the Manual Vacuum Aspiration procedure.
  Misoprostol: 400µg
- Misoprostol 200µg: Participants received misoprostol 200 µg: 1 tablet was introduced into the vagina, at least 6 hours before the Manual Vacuum Aspiration procedure.
  Misoprostol: 200µg
Period: Overall Study
Arm/Group | Misoprostol 400µg | Misoprostol 200µg
Started | 106 | 105
Completed | 106 | 105
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Misoprostol 400 µg: Misoprostol 400 µg 6 hours before Manual Vacuum Aspiration
- Misoprostol 200: Misoprostol 200 µg 6 hours before Manual Vacuum Aspiration
- Total: Total of all reporting groups
Arm/Group | Misoprostol 400 µg | Misoprostol 200 | Total
Number analyzed (Participants) | 106 | 105 | 211
Age, Continuous [Median (Full Range); unit: years] | 30 [16 to 46] | 31 [15 to 49] | 30 [15 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 105 | 211
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 29 | 26 | 55
  Brazilian indian | 0 | 1 | 1
  White | 76 | 77 | 153
  Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Brazil | 106 | 105 | 211
Obstetric history [Median (Full Range); unit: cases] — Obstetric history was assessed as the median number of previous miscarriages, median number of previous deliveries post 20 weeks gestation (para/parity), median number of previous pregnancies (gesta/gravida) AND median number of previous deliveries before 20 weeks gestation (miscarriages); all of them used the full range
  cases
    Gesta | 2 [1 to 8] | 2 [1 to 8] | 2 [1 to 8]
    Para | 1 [0 to 7] | 1 [0 to 6] | 1 [0 to 7]
    Miscarriages | 1 [1 to 7] | 1 [1 to 4] | 1 [1 to 7]
Time from misoprostol to procedure [Mean (Standard Deviation); unit: hours] | 6.38 (1.47) | 6.37 (1.28) | 6.37 (1.39)
Gestational age [Mean (Standard Deviation); unit: weeks] — weeks of pregnancy
  weeks | 7 (1.4) | 7.1 (1.5) | 7.1 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Required Cervix Dilation at Initiation of the Manual Vacuum Aspiration
Description: this outcome identifies patients that had to have a mechanical dilator for opening the cervix to perform appropriate Manual Vacuum Aspiration
Time Frame: baseline at initiation of the Manual Vacuum Aspiration
Population: Intention to Treat Population (all participants assigned to misoprostol 400µg or 200µg)
Measure: Count of Participants; unit: Participants
Groups:
- Misoprostol 400 µg: Misoprostol 400 µg 6 hours before intrauterine suction
  Misoprostol 400 µg: evaluate the required cervix dilation in the moment of the intrauterine suction
- Misoprostol 200 µg: Misoprostol 200 µg 6 hours before intrauterine suction
  Misoprostol 200 µg: evaluate the required cervix dilation in the moment of the intrauterine suction
Arm/Group | Misoprostol 400 µg | Misoprostol 200 µg
Number analyzed (Participants) | 106 | 105
Participants
  It was necessary (inadequate cervix dilation) | 4 | 16
  It was not necessary (adequate cervix dilation) | 102 | 89
Statistical Analysis 1: Comparison: Misoprostol 400 µg vs Misoprostol 200 µg; If there is a true difference in favour of the standard treatment of 10% (96% vs 86%), then 184 patients are required to be 95% sure that the upper limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) will exclude a difference in favour of the standard group of more than 25%; Test type: Non-Inferiority — 400µg of misoprostol yields a 96% cervical dilation > 8 mm. We considered 86% of the 200 µg misoprostol group as the minimal acceptable percentage. The non-inferiority margin was determined by 24.46; p = 0.025, difference between proportions — The null hypothesis: percentage of dilation with 400µg ≥ percentage of dilation with 200µg + 25% Alternative hypothesis: percentage of dilation with 400µg - 25% < percentage of dilation with 200µg; difference between percentages and 95% confidence interval; treatment difference = 25, 95% CI 1-sided [upper limit 97.5]
Statistical Analysis 2: Comparison: Misoprostol 400 µg vs Misoprostol 200 µg; Test type: Non-Inferiority — The non-inferiority margin was determined by ⅓ of the difference between the 400µg effect (96.7%), compared to the 200 µg dose (23.3%), i.e. 73.4 / 3 = 24.46%; p = 0.004, Chi-squared; Difference between proportions = 0.1146, 95% CI 2-sided [0.037 to 0.192] — The difference between both groups was 11.5% (95%CI = 3.7% to 19.2%)

2. Secondary Outcome: Number of Participants With a Presence of a Uterine Cervical Canal With ≥8 mm of Dilation
Description: This outcome measures how many mm of dilation the cervical canal has before the procedure. Cervical permeability (≥8 mm of dilation, used as a cut-off) was measured using Karman cannulas, from higher to low diameter.
Time Frame: Baseline before Manual Vacuum Aspiration procedure
Population: Intention to Treat (all patients assigned to 400mg or 200µg of misoprostol)
Measure: Count of Participants; unit: Participants
Arm/Group | Misoprostol 400 µg | Misoprostol 200 µg
Number analyzed (Participants) | 106 | 105
Participants
  Inadequate (<8 mm) | 30 | 50
  Adequate (≥8 mm) | 76 | 55

3. Other Pre Specified Outcome: Pain Score (VAS)
Description: Pain scores were assessed using a verbal analog scale (VAS), ranging from zero (no pain) to 10 (worst possible pain)
Time Frame: before Manual Vacuum Aspiration
Measure: Median (Full Range); unit: units on a scale - Verbal Analog Scale
Arm/Group | Misoprostol 400 µg | Misoprostol 200 µg
Number analyzed (Participants) | 106 | 105
units on a scale - Verbal Analog Scale | 0 [0 to 10] | 0 [0 to 10]
Statistical Analysis 1: Comparison: Misoprostol 400 µg vs Misoprostol 200 µg; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0]

ADVERSE EVENTS:
Time Frame: From the MVA procedure until 6 hours after the procedure
Groups:
- Misoprostol 400 µg: Misoprostol 400 µg 6 hours before MVA
- Misoprostol 200 µg: Misoprostol 200 µg 6 hours before MVA
Arm/Group | Misoprostol 400 µg | Misoprostol 200 µg
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/105
Other Adverse Events (participants affected / at risk) | 1/106 | 3/105
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol 400 µg (N=106) | Misoprostol 200 µg (N=105)
uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) — Grade 2 - medical intervention indicated
cervical laceration (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Cervical laceration occurred with Pozzi forceps traction. Local suture was performed without further treatment

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable. Pregnancies with less than 8 weeks had their procedures completely done with small diameter Karman cannulas

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: English version 2020 NCT02957305 (2020-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02957305/Prot_SAP_ICF_000.pdf